CLINICAL TRIAL: NCT01183130
Title: Compliance Monitoring in Real Time During Opioid Substitution Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The technology planned to be used in the study got outdated and therefore the study will not be conducted according to the initial protocol.
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Ulrich Tacke, Kuopio University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KUH5703434
Record Dates: First submitted 2010-08-09; First posted 2010-08-17 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2011-08

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; compliance monitoring; substitution treatment
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compliance monitoring in real time (Experimental): Patients get their opioid substitution medications in electronic compliance monitoring devices and send information of their medication intakes with mobile phone to the clinic every day during the two month study period.
  Interventions: Device: Compliance monitoring with electronic device
- Compliance monitoring (Active Comparator): Patients get their opioid substitution medications in electronic compliance monitoring devices. Information of their medication intakes will be reviewed during the weekly visits to the clinic.
  Interventions: Device: Compliance monitoring with electronic device

INTERVENTIONS:
Device: Compliance monitoring with electronic device — Electronic compliance monitoring with monitoring device (Pharma DDSi, Stora Enso) is used in control group (n=6) and device with mobile phone in intervention group (n=6). Patients in intervention group send every day the information of their medication intakes with the mobile phone to the clinic. This intervention is tested in pilot study (n=2-3) before the actual study begins.

SUMMARY:
The aim of the study is to examine whether electronic compliance monitoring in real time could offer some advantages compared to normal electronic monitoring in opioid substitution treatment. The investigators would also like know whether this method could enable the quick detection of possible problems in medication intakes and/or prevent the abuse or diversion of substitution medications.

ELIGIBILITY:
Inclusion Criteria:

* Opiate dependence
* Suboxone treatment
* Stable substitution medication dose

Exclusion Criteria:

* Chaotic situation in life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of treatment (Treatment Outcomes Profile TOP) | Every four weeks.
  Structured interview designed to measure the effectiveness and outcomes of opioid substitution treatment. Interview covers the last four weeks so it can be done every four weeks.

SECONDARY OUTCOMES:
Patients´opinions about the treatment. | Once when the study phase ends (after the 8 th study week).
  Questionnaire designed for this study to explore patients' opinions on the compliance monitoring and it's effect on the treatment and abuse and/or diversion of medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Tacke, MD, PhD, Study Director — Kuopio University Hospital, University of Eastern Finland